CLINICAL TRIAL: NCT06298279
Title: A Randomized Factorial Trial of Internet-delivered Cognitive Behaviour Therapy for Public Safety Personnel: Examining the Impact of Content Delivery Method
Brief Title: Assessing Social Learning and Course Delivery Timing in Internet-delivered Cognitive Behaviour Therapy for Public Safety Personnel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023-436
Record Dates: First submitted 2024-02-14; First posted 2024-03-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Factor 1: Tunneled or Personalized Course Delivery Factor 2: Standard or Enhanced Social Learning Resources Participants will be randomly assigned to one of four treatment conditions (tunneled delivery of ICBT with standard resources, tunneled delivery of ICBT with enhanced social learning resources, personalized delivery ICBT with standard resources, personalized delivery of ICBT with enhanced social learning resources)
Masking Description: Participants cannot be blinded to condition because ICBT (like other psychotherapies) cannot be both provided to and concealed from a participant. However, the difference between the four conditions (i.e., presence or absence of social learning resources, tunneled versus personalized course navigation) will be concealed from all participants. Because outcomes will be assessed via self-report questionnaire measures, outcomes assessor masking is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tunneled Delivery/Standard Resources (Experimental): In this arm, participants will be guided through the Self-Guided PSP Wellbeing Course in a predetermined order and using predetermined timing. Future lessons will "unlock" as previous lessons are completed.
  Participants receiving the standard resources will be presented with resources that are typically presented in PSPNET courses. This includes lesson slides case stories, do-it yourself guides, and frequently asked questions pages.
  Interventions: Behavioral: Tunneled Delivery; Behavioral: Standard Resources; Behavioral: Transdiagnostic Self-Guided ICBT
- Tunneled Delivery/Enhanced Social Learning Resources (Experimental): In this arm, participants will be guided through the Self-Guided PSP Wellbeing Course in a predetermined order and using predetermined timing. Future lessons will "unlock" as previous lessons are completed.
  Participants receiving the enhanced social learning resources will receive the same resources offered in the standard conditions (i.e., lesson slides, case stories, do-it-yourself guides, and frequently asked questions pages) and will also receive additional resources. Additional resources will include homework records to accompany the case stories, de-identified quotations from previous clients for each lesson, and a motivational video encouraging them to engage with the course.
  Interventions: Behavioral: Tunneled Delivery; Behavioral: Enhanced Social Learning Resources; Behavioral: Transdiagnostic Self-Guided ICBT
- Personalized Delivery/Standard Resources (Experimental): In this arm, participants will be able to navigate through the course modules in whichever order and at whatever pace they like. Participants will not have to complete one lesson in order to gain access to the following lesson.
  Participants receiving the standard resources will be presented with resources that are typically presented in the course. This includes lesson slides, case stories, do-it yourself guides, and frequently asked questions pages.
  Interventions: Behavioral: Personalized Delivery; Behavioral: Standard Resources; Behavioral: Transdiagnostic Self-Guided ICBT
- Personalized Delivery/Enhanced Social Learning Resources (Experimental): In this arm, participants will be able to navigate through the course modules in whichever order and at whatever pace they like. Participants will not have to complete one lesson in order to gain access to the following lesson.
  Participants receiving the enhanced social learning resources will receive the same resources offered in the standard conditions (i.e., lesson slides, case stories, do-it-yourself guides, and frequently asked questions pages) and will also receive additional resources. Additional resources will include homework records to accompany the case stories, de-identified quotations from previous clients for each lesson, and a motivational video encouraging them to engage with the course.
  Interventions: Behavioral: Personalized Delivery; Behavioral: Enhanced Social Learning Resources; Behavioral: Transdiagnostic Self-Guided ICBT

INTERVENTIONS:
Behavioral: Tunneled Delivery — Participants will be offered a pre-determined pathway to completing the 8-week course
  Arms: Tunneled Delivery/Enhanced Social Learning Resources; Tunneled Delivery/Standard Resources
Behavioral: Personalized Delivery — Participants will be able to complete course modules at their own pace and in the order that most interests them.
  Arms: Personalized Delivery/Enhanced Social Learning Resources; Personalized Delivery/Standard Resources
Behavioral: Standard Resources — Participants will receive the resources as typically included in the Self-Guided PSP Wellbeing Course.
  Arms: Personalized Delivery/Standard Resources; Tunneled Delivery/Standard Resources
Behavioral: Enhanced Social Learning Resources — Participants will receive additional intervention content.
  Arms: Personalized Delivery/Enhanced Social Learning Resources; Tunneled Delivery/Enhanced Social Learning Resources
Behavioral: Transdiagnostic Self-Guided ICBT — An ICBT course that is completed without the guidance of a therapist.

SUMMARY:
This study is a randomized factorial trial designed to evaluate unguided (i.e., purely self-help), transdiagnostic internet delivered cognitive behaviour therapy tailored for public safety personnel with tunneled of personalized course delivery and with or without the incorporation of social learning resources.

DETAILED DESCRIPTION:
Background---- Public Safety Personnel (PSP) are at an increased risk of developing mental disorders. PSP also face many barriers to accessing mental health services (e.g., stigma, location, time). The PSP Wellbeing Course is a transdiagnostic internet-delivered cognitive behaviour therapy (ICBT) course that has been specifically tailored to PSP. The effectiveness of the therapist-guided course and a self-guided course have both been supported. Consistent with the larger literature on self-guided ICBT, engagement with and outcomes of the self-guided PSP Wellbeing Course could be strengthened. Persuasive design describes using technology to influence human behaviour. The current study is designed to assess the impact of different timing options (i.e., tunneled vs. personalized) and increased social learning (i.e., standard versus enhanced social learning) on user experience, adherence, and outcomes in ICBT.

Methods--- Participants will be recruited via posts on the PSPNET social media platforms (i.e., Twitter and Facebook) and emails distributed by PSP organizations. Members of the PSPNET team will also reach out to contacts within PSP organizations to ask them to tell their colleagues about the proposed research. All interested participants will be directed to the study website (www.pspnet.ca) to complete an online screening questionnaire. As part of this questionnaire, they will be presented with a consent form explaining the screening. After consent is given, clients will be assessed for eligibility using an online screening questionnaire. The online screening questionnaire captures demographic information (e.g., sex, ethnicity, location), information about depression and other mental health issues, and background information (e.g., medical history, mental health history, symptoms).

After completing the questionnaires, participant responses will be reviewed by PSP staff for eligibility. Clients who are eligible will be randomized into one of four conditions. Participants who do not meet criteria, but are over the age of 18, will not be randomized and will instead be enrolled into the "treatment-as-usual" version of the course, which consists of a tunneled delivery and standard resources. Ineligible participants' data will not be included in analyses. Individuals under the age of 18 will not be eligible for any services.The two factors in the trial are:

Factor 1: Tunneled course delivery or personalized course delivery

Factor 2: Standard or enhanced social learning resources.

As this is a factorial trial with two factors, each client will be randomized to one of four conditions:

Condition 1: Tunneled Delivery and Standard Resources Condition 2: Tunneled Delivery and Enhanced Social Learning Resources Condition 3: Personalized Delivery and Standard Resources Condition 4: Personalized Delivery and Enhanced Social Learning Resources

Randomization will occur within 2 business-days of completion of the screening questionnaires.

All participants will receive the Self-Guided PSP Wellbeing Course, a transdiagnostic internet intervention. The program is an adaptation of a previous Australian course, the Wellbeing Course. The course involved 5 lessons that are typically completed over an 8 week period, though participants will have access to the course materials for up to 26 weeks. The content is focused on cognitive behavior therapy and relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills). All participants are presented with worksheets at the end of each lesson that contain exercises that facilitate skill acquisition. Participants will be sent automatic emails reminding them to stay engaged with the lessons and to complete questionnaires. Participants will complete questionnaires at screening, 4 weeks, 8 weeks (post-treatment), and 20 weeks (post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current or former public safety personnel (or public safety personnel trainee)
* Residing in Canada at time of enrollment
* Has regular access to the internet
* Confirms intent to participate in study

Exclusion Criteria:

* Not 18 years of age or older
* Not a current or former public safety personnel (or public safety personnel trainee)
* Not residing in Canada at time of enrollment
* Does not have regular access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7-item (GAD-7) | Screening, 4 weeks, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Change in total GAD-7 anxiety score which can range from 0 to 21. Higher scores indicate greater anxiety (worse outcome)
Patient Health Questionnaire-9 (PHQ-9) | Screening, 4 weeks, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Change in total PHQ-9 score which can range from 0 to 27. Higher scores indicate greater depression (worse outcome)
PTSD Checklist for the DSM-5 (PCL-5) | Screening, 4 weeks, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Change in total PCL-5 score which can range from 0 to 80. Higher scores indicate greater posttraumatic stress symptoms (worse outcome)
Engagement | From date of enrollment to 26 weeks (post-treatment)
  Internal portal recordings of participant how many lessons participants accessed, how many additional resources were accessed, and the dates of access. Greater course access is indicative of greater engagement within the course.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) | Screening, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Change in total WSAS score which can range from 0 to 40. Higher scores indicate greater levels of distress related to functional impairment (worse outcome)
Brief Resilience Scale (BRS) | Screening, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Change in total BRS score which can range from 0 to 30. Higher scores indicate greater resilience (better outcome)
Healthcare Use Questionnaire | Screening, 8 weeks (post-treatment), and 20 weeks (post-treatment)
  Bespoke questionnaire regarding access to healthcare resources
Case Story Questionnaire | 8-weeks (post-treatment)
  Bespoke questionnaire inquiring about participants' experiences with the case stories. Participants receiving enhanced social learning resources will be asked additional questions about the enhanced social learning resources.
Treatment Satisfaction Questionnaire | 8-weeks (post-treatment)
  Bespoke 7-item questionnaire assessing participants' treatment satisfaction.
Digital Behavior Change Interventions Engagement Scale (DCBI) | 8-weeks (post-treatment)
  The DBCI is a questionnaire where participants are asked to rate their feelings of engagement with online interventions, which can range from 0-56. Higher scores are indicative of more positive feelings about engagement.

OTHER OUTCOMES:
Post-treatment Semi-structured interview | 8-10 weeks (post-treatment)
  A semi-structured interview developed to assess for clients experiences within the course.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No